CLINICAL TRIAL: NCT04100135
Title: GORE® CARDIOFORM Septal Occluder Migraine Clinical Study: A Study to Evaluate the Safety and Efficacy of Transcatheter Closure of Patent Foramen Ovale for Relief of Migraine Headaches
Brief Title: GORE® CARDIOFORM Septal Occluder Migraine Clinical Study
Acronym: RELIEF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Dissatisfactory enrollment rate with no safety concerns
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GSO 17-03
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Migraine; Patent Foramen Ovale; PFO - Patent Foramen Ovale
Keywords: Migraine; PFO; Patent Foramen Ovale; Migraine aura
MeSH Terms: conditions — Migraine Disorders; Foramen Ovale, Patent; Migraine with Aura | interventions — thienopyridine; Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Test Arm (Experimental): Device PFO closure with the GORE® CARDIOFORM Septal Occluder
  Interventions: Device: Actual device PFO closure; Drug: Thienopyridine (clopidogrel or prasugrel)
- Control Arm (Sham Comparator): Sham device PFO closure (PFO not closed)
  Interventions: Drug: Thienopyridine (clopidogrel or prasugrel); Device: Sham device PFO closure

INTERVENTIONS:
Device: Actual device PFO closure — Actual PFO closure with the GORE® CARDIOFORM Septal Occluder
  Other Names: GORE® CARDIOFORM Septal Occluder
  Arms: Test Arm
Drug: Thienopyridine (clopidogrel or prasugrel) — Thienopyridine tablets (clopidogrel or prasugrel) administered for 6 months following device procedure
  Other Names: Plavix; Effient
Device: Sham device PFO closure — Sham (simulated) device PFO closure with result of no device implantation and no PFO closure
  Arms: Control Arm

SUMMARY:
Multi-center, prospective, randomized, placebo- and sham-controlled study to evaluate the GORE® CARDIOFORM Septal Occluder for migraine headache relief

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18-55 years of age at the screening visit.
2. Subject is willing and capable of complying with the study protocol requirements, including the specified follow-up period, and can be contacted by telephone.
3. Subject signed an Informed Consent Form prior to study participation.
4. Subject's symptoms meet International Classification of Headache Disorders - 3 (ICHD-3) Diagnostic Criteria for migraine with or without aura.
5. Subject has at least one year of migraine symptom duration.
6. Subject had migraine onset younger than 50 years of age.
7. Subject has more than one migraine headache day per week on average by history - headache day defined as: headache that meets ICHD-3 criteria for migraine or probable migraine with or without aura and lasts at least four hours or administration of acute medication before four hours (regardless of clinical response to acute medication).
8. Subject has tried and failed at least two preventive medications at adequate dosage for an adequate duration, in the judgement of the study site neurologist, and be from two separate classifications of the following classes of drugs: antidepressants, antihypertensive, anticonvulsant, onabotulinumtoxin A, CGRP inhibitors or other treatments with at least one positive randomized placebo-controlled trial (See APPENDIX A).
9. Subject must exhibit stable dosage on their preventive migraine medication for at least two months prior to the screening visit and agree to continue preventive medication at current dosage throughout the duration of the study.
10. Female subjects are currently not pregnant, breastfeeding or lactating and not planning pregnancy during their participation in the study.
11. Female subjects capable of becoming pregnant agree to use birth control or abstinence during their participation in the study.
12. Presence of Patent Foramen Ovale (PFO), as determined initially by positive bubble study utilizing Transthoracic Echocardiography (TTE) or transesophageal echocardiography (TEE), demonstrating right-to-left shunting.
13. Subject is willing to complete daily electronic migraine headache log.
14. Subject is not planning surgery during their participation the study.

Exclusion Criteria:

1. Subject is currently enrolled in any pre-approval investigational study. (Does not apply to long-term post-market studies unless participation might interfere clinically with the RELIEF endpoints.)
2. Subject has known organic issues which may cause headaches (e.g., temporo-mandibular joint, brain tumor, cervical spinal issues, known seizure disorder, etc.).
3. Subjects with hemicrania continua, post-traumatic headache, or other trigeminal autonomic cephalalgia secondary headache disorders.
4. Subject has known hypersensitivity or contraindication to thienopyridines.
5. Subject is currently taking a P2Y12 inhibitor (See APPENDIX B).
6. Subject has need for chronic oral anticoagulation therapy (e.g., atrial fibrillation, mechanical heart valve, etc.) (See APPENDIX B).
7. Subject has need for chronic antiplatelet therapy.
8. Subject has need for daily use of non-steroidal anti-inflammatory drugs (NSAIDs) (See APPENDIX B).
9. Subject has a history of thrombocytopenia within one year, or platelet count <100,000 mm3 identified during the screening phase.
10. Subject has severe hepatic impairment with reduced synthetic function as documented by prolongation of PT/PTT or total bilirubin > 3.0 mg/dL identified during the screening phase.
11. Subject has any history of stroke, TIA, or intracranial hemorrhage.
12. Subject has previously implanted pacemaker, IVC filter, PFO closure device, ASD closure device, left atrial appendage closure device OR any cardiac surgical or interventional history which, in the investigator's opinion, would preclude them from study participation.
13. Subject has documented right-to-left shunt source in addition to PFO, such as pulmonary arteriovenous malformation.
14. Subject used opioids, marijuana (medical or recreational) or butalbital-containing medications for acute migraine headache treatment four or more times per month on average within the past six months.
15. Subject abuses alcohol and/or drugs in the opinion of the Investigator.
16. Subject is unable to understand the study requirements or has a history of non-compliance with medical advice.
17. Subject has a history of clinically significant bleeding within six months of the screening visit, any active bleeding, or active peptic ulcer disease.
18. Subject has an uncontrolled arrhythmia or, if on therapy, within the past 90 days has evidence of arrhythmia control failure (e.g., supraventricular tachycardia while under rate control or atrial fibrillation while under rhythm control).
19. Subject has elevated pulmonary vascular resistance (PVR) which, in the opinion of the implanting physician, precludes safe defect closure.
20. Subject has uncontrolled systemic hypertension at the time of screening, in the opinion of the investigator.
21. In the opinion of the Investigator, patient has anatomic criteria identified during the screening evaluation and/or the screening echocardiogram that are unfavorable for successful placement of the GORE® CARDIOFORM Septal Occluder.
22. Subject has active infection at the time of screening that cannot be treated.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Reduction in Migraine Headache Days: mean reduction in the number of migraine headache days per month from baseline to follow-up headache days per month from baseline to follow-up | Week 40
  Primary Efficacy Endpoint
Proportion of subjects with any Serious Adverse Event (SAE) related to the study device or study procedure through 30 days post-procedure | 30 days post-procedure
  Primary Safety Endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sommer, MD, Principal Investigator — Columbia University; David Dodick, MD, Principal Investigator — Mayo Clinic
Locations (15):
- United States (15):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - UCLA Health, Los Angeles, California
  - Santa Barbara Cottage Hospital Research Institute, Santa Barbara, California
  - South Denver Cardiology, Denver, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Mercy One Iowa Heart Center, West Des Moines, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - University at Buffalo, Buffalo, New York
  - SJH Cardiology Associates, Liverpool, New York
  - Columbia University Medical Center, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - Aurora St Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No